CLINICAL TRIAL: NCT04917016
Title: B-HCG Levels in Women Undergoing Hysteroscopy for Removal of Retained Products of Conception
Brief Title: B-HCG Levels in Women Diagnosed With Retained Products of Conception
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Noam Smorgick MD, Director of Minimally Invasive Gynecologic Surgery, Assaf-Harofeh Medical Center
Other Study IDs: 0195-19-ASF
Record Dates: First submitted 2021-01-13; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Retained Products of Conception
Keywords: Hysteroscopy; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Women undergoing hysteroscopy for removal of RPOC
  Interventions: Diagnostic Test: Plasma B-HCG levels

INTERVENTIONS:
Diagnostic Test: Plasma B-HCG levels — Blood sample

SUMMARY:
Retained Products of Conception (RPOC) is a condition where gestational tissue remains in the uterus after birth or after a surgical or medical abortion. This condition may cause significant bleeding, infection, and long-term intrauterine adhesions associated with fertility problems and pregnancy complications (Asherman's syndrome). RPOC are diagnosed according to the clinical and ultrasound findings (such as an echogenic foci in the uterine cavity with Doppler blood flows). However, the diagnosis of RPOC by clinic and ultrasound characteristics is inaccurate and false positive results are reported in up to 40% of women undergoing a surgical procedure for RPOC removal (most often by hysterosocpy). However, surgery also carries a risk of complications and intrauterine infections. Therefore, the need arises for additional tools to improve the diagnosis available today in order to minimize the need for surgical procedures as much as possible.

The production and secretion of the B-HCG occurs in the placenta and begins after blastocyst implantation. The B-HCG levels increase in other placental pathologies such as gestational trophoblastic disease (GTD). Accordingly, the investigators hypothesized that in cases of placental remnants a secretion of B-HCG may be detected and quantified.

In this prospective, non-interventional study the investigators' aim is to examine whether B-HCG can be used as a marker for detecting placental remnants, compared to the currently accepted sonographic method. For this purpose, the investigators will examine the levels of B-HCG in participants undergoing hysteroscopy for removal of RPOC.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Admitted for hysteroscopy for RPOC removal following delivery
* Admitted for hysteroscopy for RPOC removal following abortion.

Exclusion Criteria:

* Low suspicion of RPOC by clinical or ultrasound examination.
* No pathology specimen available.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women >18 years admitted for hysteroscopy for RPOC removal following delivery of abortion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
B-HCG levels | From randomization to the day of surgery, assessed up to 3 months
  Plasma levels of B-HCG measured in mU/mL in women undergoing hysteroscopy for removal of RPOC

CONTACTS AND LOCATIONS:
Overall Officials: Noam Smorgick, MD Msc, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Result] Barel O, Krakov A, Pansky M, Vaknin Z, Halperin R, Smorgick N. Intrauterine adhesions after hysteroscopic treatment for retained products of conception: what are the risk factors? Fertil Steril. 2015 Mar;103(3):775-9. doi: 10.1016/j.fertnstert.2014.11.016. Epub 2014 Dec 17. PMID 25527235
- [Result] Smorgick N, Barel O, Fuchs N, Ben-Ami I, Pansky M, Vaknin Z. Hysteroscopic management of retained products of conception: meta-analysis and literature review. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:19-22. doi: 10.1016/j.ejogrb.2013.11.020. Epub 2013 Dec 1. PMID 24332096
- [Result] Smorgick N, Krakov A, Maymon R, Betser M, Tovbin J, Pansky M. Postpartum Retained Products of Conception: A Novel Approach to Follow-Up and Early Diagnosis. Ultraschall Med. 2018 Dec;39(6):643-649. doi: 10.1055/s-0043-113817. Epub 2017 Sep 21. PMID 28934813
- [Result] van den Bosch T, Daemen A, Van Schoubroeck D, Pochet N, De Moor B, Timmerman D. Occurrence and outcome of residual trophoblastic tissue: a prospective study. J Ultrasound Med. 2008 Mar;27(3):357-61. doi: 10.7863/jum.2008.27.3.357. PMID 18314513